CLINICAL TRIAL: NCT02361775
Title: Ultrasound Guided Paravertebral Catheter Versus Patient Controlled Analgesia for Postoperative Pain Control in Video Assisted Thoracoscopic Surgery: A Prospective Outcomes Study
Brief Title: Paravertebral Catheters for VATS Procedures
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1201M09227
Record Dates: First submitted 2015-02-03; First posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paravertebral catheter (Experimental): a paravertebral catheter is placed and an elastomeric pump is connected to infuse 0.2% ropivacaine postoperatively
  Interventions: Device: Paravertebral catheter; Drug: Ropivacaine; Device: Elastomeric Pump
- IV PCA (Active Comparator): opioid PCA consisting of hydromorphone is connected to patient in the post anesthesia care unit
  Interventions: Device: opioid iv pca

INTERVENTIONS:
Device: Paravertebral catheter — A catheter is placed ultrasound guided at the T5 paravertebral level
  Arms: Paravertebral catheter
Device: opioid iv pca — opioid pca consisting of hydromorphone
  Arms: IV PCA
Drug: Ropivacaine — 0.2% ropivacaine infused through paravertebral catheter
  Other Names: Naropin
  Arms: Paravertebral catheter
Device: Elastomeric Pump — Elastomeric pump connected to paravertebral catheter
  Other Names: On Q
  Arms: Paravertebral catheter

SUMMARY:
Level I randomized prospective outcomes study comparing two groups of patients. One group will receive Dilaudid patient controlled analgesia (PCA) post-operatively. The other will receive an ultrasound guided paravertebral block with indwelling paravertebral catheter with an infusion of 0.2% Ropivicaine post-operatively and a PCA.

DETAILED DESCRIPTION:
Design: Level I randomized prospective outcomes study comparing two groups of patients. One group will receive Dilaudid patient controlled analgesia (PCA) post-operatively. The other will receive an ultrasound guided paravertebral block with indwelling paravertebral catheter with an infusion of 0.2% Ropivicaine post-operatively and a PCA.

Sample Size: 50 patients Study Duration: Approximately 24 months Population:. Patients presenting to the University of Minnesota Medical Center for elective Video Assisted Thoracoscopic Surgery (VATS), for thoracic, lung, or mediastinal lesions or masses.

Primary Objective: To determine if post-operative paravertebral catheters in patients with elective VATS procedures result in decreased pain compared to patients treated with PCA for post-operative pain.

Secondary Objectives:

1. To determine whether the use of paravertebral catheters impacts the length of ICU and hospital stay for patients, compared to a PCA in patients undergoing elective Video Assisted Thoracoscopic Surgery (VATS).
2. To determine whether the use of paravertebral catheters leads to lower risk of complications, compared to use of a PCA in patients undergoing elective Video Assisted Thoracoscopic Surgery (VATS).

2. Synopsis and Medical Application:

Specific Aims:

Primary Hypothesis: Paravertebral catheters will result in improved pain control relative to PCA for post-operative pain from thoracic surgery.

Secondary Hypothesis: Paravertebral catheters will result in fewer hospital days and improved subjective respiratory function compared to patients in the PCA group.

ELIGIBILITY:
Inclusion Criteria:

* • All patients undergoing elective VATS.

Exclusion Criteria:

* • Previous difficult airway or multiple previous intubations

  * History of myasthenic syndrome
  * Systemic infection
  * Pre-existing sensory deficit
  * PT >14 or PTT >40 sec
  * Platelet count less than 50,000
  * Creatinine > 1.5
  * Allergy to local anesthetics
  * Patients who remain intubated for one week after surgery or who are unable to provide information as to their feelings of pain post-operatively for the first week post-operatively
  * Use of a spinal or epidural anesthetic for surgery
  * Daily use of opioid for more than a week
  * Lack of patient cooperation
  * Contraindication to regional anesthesia

    * Infection at injection site
    * Inability to guarantee sterile equipment or sterile conditions for the block
    * Patient refusal
    * Risk of local anesthetic toxicity
    * Coagulopathy or bleeding disorder
    * Severe respiratory disease (where the patient depends on intercostal muscle function for ventilation);
    * Ipsilateral diaphragmatic paresis;
    * Severe spinal deformities (kyphosis or scoliosis)
    * Previous thoracotomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Maximum NRS Pain score | 0-24 hours after surgery
  pain at movement or maximum in first 24 hours after surgery

SECONDARY OUTCOMES:
total opioid use | the first 5 days after surgery
  total opioids converted to morphine equivalents
length of stay | time until patient is ready to be discharged or is discharged, expected 5 days
  participants will be followed for duration of stay expected 5 days

OTHER OUTCOMES:
the number of patients with presence of nausea and vomiting | the first 5 days postoperatively
  the number of patients who have nausea and or vomiting.